CLINICAL TRIAL: NCT02082925
Title: Self-perception of Dyspnea Threshold During the 6-minute Walk Test (DT6): A New Tool for Individualized Exercise Training With Chronic Obstructive Pulmonary Disease Patients (COPD)
Brief Title: Dyspnea Threshold During 6 Minutes Walk Test
Acronym: SD6
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 5 Santé (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FVIE_SD6
Record Dates: First submitted 2014-03-04; First posted 2014-03-10 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-03

CONDITIONS: COPD
Keywords: Exercise training; Dyspnea threshold; 6MWT
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- COPD patient (Experimental)
  Interventions: Other: Patient has to get up his hand when he defined his dyspnea threshold during 6MWT

INTERVENTIONS:
Other: Patient has to get up his hand when he defined his dyspnea threshold during 6MWT

SUMMARY:
In view of the multiple limitations and restrictions relative to CPET (technical, time, physical…), determination of individualized training threshold from this evaluation is today not possible for a lot of patients.

The aim of this study was to propose a new clinical tool from 6MWT for individualized exercise training: the dyspnea threshold (DT6).

ELIGIBILITY:
Inclusion Criteria:

* COPD
* with or without rest and/or ambulation oxygen therapy

Exclusion Criteria:

* exacerbation in the previous four weeks
* with a restrictive or mixed respiratory syndrome, angina , recent heart attack (< 1 month) or coronary progressive pathology
* under beta-blockers
* cognitive or motor problems which limit significantly comprehension or achievement of evaluations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change of heart rate between 1st and 2nd 6MWT | at baseline (2 days after entry in pulmonary rehabilitation)

SECONDARY OUTCOMES:
Change of heart rate between VT (CPET) and DT6 (6MWT) | At baseline

CONTACTS AND LOCATIONS:
Overall Officials: Nelly HERAUD, Study Director
Locations (1):
- Clinique du Souffle La Vallonie, Lodève, France